CLINICAL TRIAL: NCT07015515
Title: Acute Effects of Push-Up Exercise Performed Under Varying Blood Flow Restriction Conditions on Upper Extremity Explosive Power Performance
Brief Title: PAPE Effect With Blood Flow Restriction and Push-Up Exercise (Post-Activation Performance Enhancement)
Acronym: PAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Şensu Dinçer, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PAPE-BFR-2025
Record Dates: First submitted 2025-05-30; First posted 2025-06-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Blood Flow Restriction Exercise
Keywords: BFR; push-up exercise; PAPE; radar measurement; explosive power
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blood flow restriction exercise group (Experimental): Participants will perform push-up exercises with 50% arterial occlusion pressure applied to their dominant arm. The cuff is inflated before the exercise and maintained throughout 3 sets of 5 repetitions. There is a 2-minute rest between sets.
  Interventions: Other: Blood flow restriction exercise group
- Sham Blood flow restriction exercise group (Placebo Comparator): In this group, a BFR cuff will be placed on the upper extremity in the same location as in the real BFR group. During the application, the participant will be led to believe that the cuff is being inflated, although no actual pressure will be applied. The participant will see the cuff being wrapped and apparently inflated, but there will be no physical pressure restricting circulation during the exercise. This aims to control the psychological effects (e.g., the belief that "something is being applied") on performance.
  Interventions: Other: Sham blood flow restriction exercise
- Control group (Active Comparator): Participants perform push-up exercises without any cuff application. The same repetition and rest protocol is followed.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Sham blood flow restriction exercise — a BFR cuff will be placed on the upper extremity in the same location as in the real BFR group. During the application, the participant will be led to believe that the cuff is being inflated, although no actual pressure will be applied. The participant will see the cuff being wrapped and apparently inflated, but there will be no physical pressure restricting circulation during the exercise. This aims to control the psychological effects (e.g., the belief that "something is being applied") on performance
  Arms: Sham Blood flow restriction exercise group
Other: Control group — Participants perform push-up exercises without any cuff application. The same repetition and rest protocol is followed
  Arms: Control group
Other: Blood flow restriction exercise group — Participants will perform push-up exercises with 50% arterial occlusion pressure applied to their dominant arm. The cuff is inflated before the exercise and maintained throughout 3 sets of 5 repetitions. There is a 2-minute rest between sets.
  Arms: Blood flow restriction exercise group

SUMMARY:
This study aims to compare the acute effects of push-up exercises performed under different blood flow restriction (BFR) conditions on upper extremity explosive strength performance, measured via the seated unilateral medicine ball throw test.

DETAILED DESCRIPTION:
The study includes three push-up conditions (BFR, sham BFR, and no BFR). Performance is evaluated via medicine ball throws at the 4th, 8th, and 12th minutes post-exercise. Exercises are applied in a crossover design with 50% limb occlusion pressure (LOP) BFR, sham, and control arms. Throw distance and ball velocity (measured by radar device) are primary outcomes. RPE scale is used to assess perceived exertion.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 25 years old
* Being a volleyball player
* Having trained regularly in the last 6 months
* Ability to perform at least 5 repetitions of push-up with own body weight
* Voluntarily agreeing to participate and signing the informed consent form

Exclusion Criteria:

* History of shoulder or upper extremity injury requiring physical therapy or surgery
* History of venous thromboembolism
* Hematological disorders
* Coronary artery disease
* Peripheral arterial disease
* Hypertension (systolic/diastolic > 140 mmHg/90 mmHg)
* History or high risk of deep vein thrombosis
* Blood clotting disorders
* Poor circulation
* Inadequate lymphatic system
* History of endothelial dysfunction
* Varicose veins
* Peripheral vascular disease
* Diabetes
* Easy bruising
* Active infection
* Cancer
* Renal failure
* Pregnancy
* Intolerance to intervention

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
throw distance | will be measured immediately after the exercise protocol is completed three times at 4th, 8th, and 12th minutes
  Seated unilateral medicine ball throw distance (in cm) -

SECONDARY OUTCOMES:
Ball velocity (km/h) | will be measured by radar device after completion of the exercise three times at 4th, 8th, and 12th minutes
  speed at which a ball travels immediately after being thrown
Rating of Perceived Exertion (RPE) | 1 day (will be assessed at the end of the push-up exercise)
  will be assessed via Borg Rating of Perceived Exertion Scale (6-20). Borg scale is used o quantify an individual's subjective perception of exercise intensity. It provides a numerical scale, typically ranging from 6 to 20. Higher scores on the scale indicate a greater subjective sense of difficulty or effort perceived by the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Şensu Dinçer, Principal Investigator — Istanbul University
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)